CLINICAL TRIAL: NCT03988634
Title: A Multicenter, Randomized, Double-blind, Double Dummy, Parallel Group, Active-controlled Study to Evaluate the Effect of Sacubitril/Valsartan (LCZ696) Versus Valsartan on Changes in NT-proBNP, Safety, and Tolerability in HFpEF Patients With a WHF Event (HFpEF Decompensation) Who Have Been Stabilized and Initiated at the Time of or Within 30 Days Post-decompensation (PARAGLIDE-HF)
Brief Title: Changes in NT-proBNP, Safety, and Tolerability in HFpEF Patients With a WHF Event (HFpEF Decompensation) Who Have Been Stabilized and Initiated at the Time of or Within 30 Days Post-decompensation (PARAGLIDE-HF)
Acronym: PARAGLIDE-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696DUS01
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Heart failure with preserved ejection fraction (HFpEF); Heart failure hospitalization; NYHA; NT-proBNP; Acute decompensated heart failure; Sacubitril/valsartan; Global evaluation of treatment effectiveness (GETE); Worsening Heart Failure
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan; sacubitril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sacubitril/valsartan (LCZ696) (Experimental): Study treatment was titrated to the target dose of sacubitril/valsartan (LCZ696) 97/103 mg twice daily (Dose Level 3).
  Patients were required to take a total of two tablets twice daily (one tablet of active sacubitril and valsartan , and one tablet of valsartan matching placebo)
  Interventions: Drug: sacubitril/valsartan; Drug: valsartan matching placebo
- valsartan (Active Comparator): Study treatment was titrated to the target dose of valsartan 160 mg twice daily (Dose Level 3).
  Patients were required to take a total of two tablets twice daily (one tablet of active valsartan, and one tablet of sacubitril and valsartan matching placebo)
  Interventions: Drug: valsartan; Drug: sacubitril/valsartan matching placebo

INTERVENTIONS:
Drug: sacubitril/valsartan — Sacubitril/valsartan (LCZ696) was available as 24/26 mg, 49/51 mg, and 97/103 mg in tablet form to be taken orally, twice daily
  Other Names: LCZ696
  Arms: sacubitril/valsartan (LCZ696)
Drug: valsartan — Valsartan was available as 40 mg, 80 mg, and 160 mg in tablet form to be taken orally, twice daily
  Arms: valsartan
Drug: sacubitril/valsartan matching placebo — Sacubitril/valsartan (LCZ696) matching placebo was available as tablet form to be taken orally, twice daily
  Arms: valsartan
Drug: valsartan matching placebo — Valsartan matching placebo was available as tablet form to be taken orally, twice daily
  Arms: sacubitril/valsartan (LCZ696)

SUMMARY:
The effect of sacubitril/valsartan vs. valsartan on changes in NT-proBNP, safety, and tolerability in HFpEF patients with a WHF event (HFpEF decompensation) who had been stabilized and initiated at the time of or within 30 days post-decompensation.

DETAILED DESCRIPTION:
This study used a randomized, double-blind, double-dummy, active-controlled, parallel group design conducted across 100 centers in the US and Canada. The study duration was a maximum of 20 months (minimum follow up was 8 weeks).

Randomized patients were deemed hemodynamically stabilized and needed to meet all inclusion and none of the exclusion criteria. Patients were randomized 1:1 to LCZ696 or valsartan. Initial dose at randomization was determined based on the patient's previous dose of or lack of ACEi/angiotensin receptor blocker (ARB) immediately prior to current worsening heart failure (WHF) event (heart failure with preserved ejection fraction [HFpEF]) decompensation, or at the time of post-decompensation randomization.

LCZ696 dose or valsartan dose levels may have been increased to the targeted desired dose of 97/103 mg [200 mg] BID or valsartan 160 mg BID on an every 2-week basis or earlier based on clinical need and investigator judgment. Every effort was made to titrate to and maintain patients on the target dose level, as tolerated by the patient.

To maintain the blinding, patients were required to take their assigned active treatment tablet along with placebo matching the opposite treatment BID.

The protocol had 4 amendments. Protocol Version 00 (Original Protocol) included a double-blind phase through Week 8 followed by an open-label phase during Weeks 8 to 12. Protocol Amendment 01 omitted the open-label phase and followed patients for a maximum of 20 months in a double-blinded treatment phase. Throughout all protocol versions, the primary endpoint remained the time-averaged proportional change in N-terminal pro-brain natriuretic peptide (NT-proBNP) from Baseline to Weeks 4 and 8. The most recent protocol amendment (Amendment 04) reduced the sample size to approximately 450 patients (from 800) with 85% power for the primary endpoint, deemphasizing the statistical power for key secondary clinical endpoints; however, clinical events were still assessed as secondary endpoints.

No efficacy analyses include "OPEN LABEL' data. After Protocol Amendment 01, the open-label option was removed from the study, only the 233 patients randomized in the Double-blind Phase Sacubitril+ Valsartan (LCZ696) and the 233 patients randomized in the Double-blind Phase Valsartan arms were included in the efficacy analysis.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Signed informed consent must be obtained prior to participation in the study
2. Patients >=18 years of age, male or female
3. Current hospitalization for Worsening Heart Failure (WHF) (HFpEF decompensation), or within 30 days of discharge following a WHF event (defined as hospitalization, emergency department (ED) visit or out-of-hospital urgent HF visit, all requiring IV diuretics). Patients with a diagnosis of acute heart failure had to have symptoms and signs of fluid overload (i.e. jugular venous distention, edema or rales on auscultation or pulmonary congestion on chest x-ray). Eligible patients were randomized after IV diuresis for HFpEF is given (and no earlier than 36 hours from their last ACEi dose if applicable) and within 30 days post-decompensation after presentation with acute HFpEF decompensation and meeting the following definitions of hemodynamic stability:

   Randomized patients were hemodynamically stable defined in this study as:
   1. SBP >=100mmHg for the preceding 6 hours prior to randomization; no symptomatic hypotension
   2. No increase (intensification) in IV diuretic dose within last 6 hours prior to randomization
   3. No IV inotropic drugs for 24 hours prior to randomization
   4. No IV vasodilators including nitrates within last 6 hours prior to randomization
4. HFpEF with most recent LVEF > 40% (within past 3 months)
5. Elevated NT-proBNP or BNP at the time of acute HFpEF decompensation or post-decompensation screening (and within 72 hours for out-of-hospital randomization, if applicable):

   1. Patients not in Atrial Fibrillation(AF) at the time of biomarker assessment: NT-proBNP >= 500pg/mL or BNP >= 150 pg/mL; patients in AF at the time of biomarker assessment: NT-proBNP >= 1000pg/mL or BNP >= 300 pg/mL
   2. Patients recruited in-hospital were randomized based on the qualifying local lab value in-hospital NT-proBNP or BNP value.
   3. Patients enrolled post-decompensation can be randomized based on their NT-proBNP or BNP value in the following way:

   i. if enrolling in post-decompensation setting then need eligible screening/local NTproBNP/BNP within 72 hours of randomization. The test value could be from recent hospitalization if within 72 hours or ii. would require (re)drawing NT-proBNP or BNP labs in post-decompensation setting if the lab value is not already available within the last 72 hours).

6) Has not taken an ACEi for 36 hours prior to randomization

EXCLUSION CRITERIA:

1. Any clinical event within the 90 days prior to randomization that could have reduced the LVEF (i.e., myocardial infarction (MI), coronary artery bypass graft (CABG), unless an echo measurement was performed after the event confirming the LVEF to be > 40%
2. Entresto™ (sacubitril/valsartan) usage within the past 60 days
3. eGFR < 20ml/min/1.73 m2 as measured by the simplified Modification of Diet in Renal Disease (MDRD) formula at most recent assessment prior to randomization and within 24 hours prior to inpatient randomization or 72 hours prior to outpatient randomization
4. Serum potassium > 5.2 mEq/L at most recent assessment prior to randomization and within 24 hours prior to inpatient randomization or 72 hours prior to outpatient randomization
5. Acute coronary syndrome, stroke, transient ischemic attack; cardiac, carotid or other major CV surgery; percutaneous coronary intervention (PCI) or carotid angioplasty, within 30 days prior to randomization
6. Probable alternative diagnoses that in the opinion of the investigator could account for the patient's HF symptoms (i.e. dyspnea, fatigue) such as significant pulmonary disease (including primary pulmonary HTN), anemia or obesity.
7. Isolated right HF in the absence of left-sided structural heart disease
8. History of hypersensitivity (i.e. including angioedema), known or suspected contraindications, or intolerance to any of the study drugs including ARNIs (i.e. sacubitril/valsartan), and/or ARBs
9. Patients with a known history of angioedema due to any etiology
10. Patients with a history of heart transplant or LVAD, currently on the transplant list, or with planned intent to implant LVAD or CRT device within the initial three months of enrollment during the trial
11. A cardiac or non-cardiac medical condition other than HF with an estimated life expectancy of < 6 months
12. Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy including suspected or confirmed amyloid heart disease (amyloidosis)
13. Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or flutter with a resting ventricular rate > 110 bpm
14. Clinically significant congenital heart disease felt to be the cause of the patient's symptoms and signs of HF
15. Coronary or carotid artery disease or valvular heart disease likely to require surgical or percutaneous intervention within the duration of the trial
16. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
17. Known hepatic impairment (as evidenced by total bilirubin > 3 mg/dL, or increased ammonia levels, if performed), or history of cirrhosis with evidence of portal hypertension such as varices
18. Participation in any other clinical trial involving investigational agents or devices within the past 30 days
19. Current confirmed COVID19 infection
20. Past COVID19 infection with persistent symptom burden suspected due to COVID19 (further defined in Section 5.2).
21. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
22. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of investigational drug and for 7 days off of study drug. Highly effective contraception methods are defined in protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (95):
- United States (87):
  - University of Calif Irvine Med Cntr, Irvine, California
  - Memorial Care Health System Memorialcare Long Beach, Long Beach, California
  - University Of Southern California ., Los Angeles, California
  - University Of Southern California, Los Angeles, California
  - San Diego Cardiac Center, San Diego, California
  - Zuckerberg General W84 Research ., San Francisco, California
  - Sutter Health Network ., San Pablo, California
  - Helping Hands Medical Associates INC, Santa Ana, California
  - St Francis Medical Center, Colorado Springs, Colorado
  - Colorado Heart and Vascular ., Lakewood, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Hartford Healthcare Headache Center, West Hartford, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Cardiology Physicians PA ., Newark, Delaware
  - University of Florida Health ., Gainesville, Florida
  - New Generation of Medical Research Avera Health N Central Heart, Hialeah, Florida
  - University of Florida Health Science Center, Jacksonville, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Morehouse School Of Medicine, Atlanta, Georgia
  - Emory University School of Medicine/Winship Cancer Institute, Atlanta, Georgia
  - University Cardiology Associates, Augusta, Georgia
  - St Lukes Idaho Cardiology Associates CLCZ696BUS13, Boise, Idaho
  - University of Chicago ., Chicago, Illinois
  - Amita Health, Elk Grove Village, Illinois
  - Midwest Cardiovascular Institute ., Oakbrook Terrace, Illinois
  - Advocate Medical Group ., Park Ridge, Illinois
  - Unity Point Health Methodist, Peoria, Illinois
  - OSF HealthCare, Peoria, Illinois
  - Northwestern Medicine Northwestern University, Winfield, Illinois
  - Midwest Cardiovascular Research and Education Foundation ., Elkhart, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - Franciscan Health Services Research Center ., Indianapolis, Indiana
  - Indiana University Health, Muncie, Indiana
  - Reid Hosp And Hlth Care Services, Richmond, Indiana
  - The Uni of Kansas Medical Center, Kansas City, Kansas
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - The Franciscan Missionaries, Baton Rouge, Louisiana
  - Northern Light Easter Maine Medical Center ., Bangor, Maine
  - Johns Hopkins Univ School of Med, Baltimore, Maryland
  - Tidal Health Peninsula Regional Inc ., Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Univeristy Medical Center ., Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr CLCZ696D2301, Boston, Massachusetts
  - University of Michigan Hs, Ann Arbor, Michigan
  - Detroit Medical Center Cardiovascular Clinical Trial ., Detroit, Michigan
  - Henry Ford Hospital Cardiovascular Medicine, Detroit, Michigan
  - Trinity Health Michigan Heart ., Ypsilanti, Michigan
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Nebraska Heart Institute CHI Health Nebraska, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Univ Medical Center Las Vegas, Las Vegas, Nevada
  - R Ins For Heart And Vascular Health, Reno, Nevada
  - Inspira Health Network, Elmer, New Jersey
  - Cooper University Health Care, Haddon Heights, New Jersey
  - Saint Michael Medical Center, Newark, New Jersey
  - Cedar Multi-Specialty Clinic, Albuquerque, New Mexico
  - Albany Associates In Cardiology, Albany, New York
  - New York Presbyterian Queens ., Flushing, New York
  - United Health Services Office Of Clinical Trails CLCZ696BUS01, Johnson, New York
  - Northwell Health ., Manhasset, New York
  - Mount Sinai Hospital ., New York, New York
  - HealthQuest, Poughkeepsie, New York
  - Catholic Hlth Svcs of Long Island, Roslyn, New York
  - Mount Sinai Health System, Staten Island, New York
  - Stony Brook University Medical Center CLCZ696G2301, Stony Brook, New York
  - Montefiore Medical Center ., The Bronx, New York
  - University Of North Carolina At Chapel Hill CRLX030A2209, Chapel Hill, North Carolina
  - Duke Health, Durham, North Carolina
  - Cleveland Clinic Foundation ., Cleveland, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - St John Health System, Bartlesville, Oklahoma
  - Regional Medical Labaratory, Tulsa, Oklahoma
  - Jefferson Abington ., Abington, Pennsylvania
  - Allegheny Valley Hospital ., Natrona Heights, Pennsylvania
  - Capital Area Research LLC CACZ885M2301, Newport, Pennsylvania
  - Thomas Jefferson Univ Hospital ., Philadelphia, Pennsylvania
  - Regional Health Clinic Research ., Rapid City, South Dakota
  - North Central Heart ., Sioux Falls, South Dakota
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
  - Pharma Tex Research ., Amarillo, Texas
  - Baylor University Medical Center ., Dallas, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - The University of Vermont Medical Center CRLX030A2301, Burlington, Vermont
  - Centra Health, Lynchburg, Virginia
  - Swedish Medical Ctr Cardiovascular Re, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health CLCZ696BUS01, Madison, Wisconsin
- Canada (8):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saguenay, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of the patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Peters AE, Li S, Cyr D, Williamson KM, Zieroth S, Fudim M, Ward JH, Mentz RJ. Influence of ejection fraction on outcomes with sacubitril/valsartan in patients with worsening heart failure with EF>40%: The PARAGLIDE-HF Trial. Am Heart J. 2025 Nov;289:158-167. doi: 10.1016/j.ahj.2025.04.023. Epub 2025 Apr 21. PMID 40268180
- [Derived] Rambarat P, Erickson T, Cyr D, Ward J, Hernandez A, Morrow D, Starling R, Velazquez E, Zieroth S, Williamson K, Solomon S, Mentz R. Effects of angiotensin-neprilysin inhibition in women vs men: Insights from PARAGLIDE-HF. Am Heart J. 2025 Oct;288:41-51. doi: 10.1016/j.ahj.2025.03.017. Epub 2025 Mar 31. PMID 40174692
- [Derived] Shoji S, Cyr DD, Hernandez AF, Velazquez EJ, Ward JH, Williamson KM, Sarwat S, Starling RC, Desai AS, Zieroth S, Solomon SD, Mentz RJ. Win Ratio Analyses Using a Modified Hierarchical Composite Outcome: Insights From PARAGLIDE-HF. Am Heart J. 2025 Feb;280:70-78. doi: 10.1016/j.ahj.2024.10.020. Epub 2024 Nov 4. PMID 39505123
- [Derived] Fudim M, Cyr DD, Ward JH, Hernandez AF, Lepage S, Morrow DA, Sharma K, Claggett BL, Starling RC, Velazquez EJ, Williamson KM, Desai AS, Zieroth S, Solomon SD, Braunwald E, Mentz RJ; PARAGLIDE-HF investigators. Association of Sacubitril/Valsartan vs Valsartan With Blood Pressure Changes and Symptomatic Hypotension: the PARAGLIDE-HF Trial. J Card Fail. 2024 Dec;30(12):1568-1577. doi: 10.1016/j.cardfail.2024.04.030. Epub 2024 May 26. PMID 38802053
- [Derived] Morrow DA, Velazquez EJ, Desai AS, DeVore AD, Lepage S, Park JG, Sharma K, Solomon SD, Starling RC, Ward JH, Williamson KM, Zieroth S, Hernandez AF, Mentz RJ, Braunwald E. Sacubitril/Valsartan in Patients Hospitalized With Decompensated Heart Failure. J Am Coll Cardiol. 2024 Mar 26;83(12):1123-1132. doi: 10.1016/j.jacc.2024.01.027. PMID 38508844
- [Derived] Mentz RJ, Ward JH, Hernandez AF, Lepage S, Morrow DA, Sarwat S, Sharma K, Starling RC, Velazquez EJ, Williamson KM, Desai AS, Zieroth S, Solomon SD, Braunwald E; PARAGLIDE-HF Investigators. Angiotensin-Neprilysin Inhibition in Patients With Mildly Reduced or Preserved Ejection Fraction and Worsening Heart Failure. J Am Coll Cardiol. 2023 Jul 4;82(1):1-12. doi: 10.1016/j.jacc.2023.04.019. Epub 2023 May 21. PMID 37212758
- See also: A Plain Language Trial Summary is available at www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 586 patients screened for the study, 467 patients were randomized to receive treatment, and 466 randomized patients were treated. The study had 90 sites in the US and 10 sites in Canada
Pre-assignment Details: Patients were randomized 1:1 to sacubitril/valsartan or valsartan. Randomized patients were deemed hemodynamically stabilized and needed to meet all inclusion and none of the exclusion criteria. At the randomization visit, all eligible patients were randomized via interactive response technology to one of the treatment arms.
Groups:
- Double-blind Phase Sacubitril+ Valsartan (LCZ696): Study treatment was titrated to the target dose of sacubitril/valsartan (LCZ696) 97/103 mg twice daily (Dose Level 3).
- Double-blind Phase Valsartan: Study treatment was titrated to the target dose of valsartan 160 mg twice daily (Dose Level 3).
- Open-label Phase Sacubitril+ Valsartan: Participants recruited under Protocol Version 00 (Original Protocol) and who had completed the double-blind phase before protocol amendment 01 was released. Participants were in the open-label phase from Week 8 to Week 12.
Period: Double-Blind
Arm/Group | Double-blind Phase Sacubitril+ Valsartan (LCZ696) | Double-blind Phase Valsartan | Open-label Phase Sacubitril+ Valsartan
Started (Randomized) | 234 | 233 | 0
Treated Patients | 233 | 233 | 0
Completed | 173 | 182 | 0
Not Completed | 61 | 51 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Death | 18 | 26 | 0
Not completed — Lost to Follow-up | 6 | 7 | 0
Not completed — Physician Decision | 9 | 5 | 0
Not completed — Subject decision | 24 | 13 | 0
Period: Open-Label
Arm/Group | Double-blind Phase Sacubitril+ Valsartan (LCZ696) | Double-blind Phase Valsartan | Open-label Phase Sacubitril+ Valsartan
Started (Started open label phase under Protocol Version 00) | 0 | 0 | 50
Completed | 0 | 0 | 41
Not Completed | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Technical problems | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are based on the full analysis set (FAS), as primary and secondary analysis are based on the FAS.
  The FAS consisted of all patients to whom study treatment was assigned by randomization and at least 1 dose of study treatment received.
Groups:
- Sacubitril/Valsartan (LCZ696): Study treatment was titrated to the target dose of sacubitril/valsartan (LCZ696) 97/103 mg twice daily (Dose Level 3).
- Valsartan: Study treatment was titrated to the target dose of valsartan 160 mg twice daily (Dose Level 3).
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Total
Number analyzed (Participants) | 233 | 233 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (11.95) | 70.5 (11.56) | 69.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 121 | 242
  Male | 112 | 112 | 224
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 176 | 176 | 352
  Black | 50 | 52 | 102
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  American Indian or Alaska Native | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time-averaged Proportional Change in NT proBNP From Baseline to Weeks 4 and 8
Description: To demonstrate the effect of sacubitril/valsartan vs. valsartan on time-averaged proportional change in N-terminal pro-brain natriuretic peptide (NT-proBNP) from baseline to weeks 4 and 8 in heart failure with preserved ejection fraction (HFpEF) patients with a worsening heart failure event (HFpEF decompensation) who have been stabilized for and initiated at the time of or within 30 days post-decompensation.
  Plasma NT-proBNP (pg/mL) values were averaged from Week 4 and Week 8 visits. The change from baseline to average of Week 4 and Week 8 was expressed as the geometric mean of the ratio: Week - 8/Baseline.
  NT-proBNP is a protein produced in large amounts by the heart when it is not working properly, as in heart failure.
  Baseline value was the last non-missing assessment of plasma NT-proBNP before the first administration of study drug.
Time Frame: Baseline, Average of Week 4 and Week 8
Population: Full analysis set: All patients to whom study treatment was assigned by randomization and at least 1 dose of study treatment was received. Patients with missing baseline NT-proBNP and/or missing data from both Weeks 4 and 8 were not included in the primary analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Ratio
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan
Number analyzed (Participants) | 180 | 197
Geometric Mean Ratio | 0.7200 [0.6430 to 0.8062] | 0.8425 [0.7561 to 0.9387]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Test type: Superiority; p = 0.0492, ANCOVA; Geometric Mean Ratio = 0.8546, 95% CI 2-sided [0.7307 to 0.9994] — Geometric Mean Ratio: sac/val vs valsartan

2. Secondary Outcome: Number of Pairwise Comparisons With Wins or Ties in the Endpoint Adjudication Committee (EAC)-Adjudicated Composite Hierarchical Outcome
Description: This hierarchical composite endpoint consists of 4 ordered components: 1. Time to CV death, 2. Number and times of HF hospitalizations during follow-up, 3. Number and times of urgent HF visits during follow-up, 4. Time averaged proportional change in NT-proBNP from baseline to Weeks 4 and 8. This endpoint was analyzed estimating the unmatched win ratio by comparing every participant in the sacubitril/valsartan arm to every participant in the valsartan arm to determine a winner (unmatched pairing method). For every pair, a patient is labelled a 'winner' (i.e. achieve a better clinical outcome) or a 'loser'. Otherwise they are considered tied. The reported unit is the total "wins" or "ties" for each treatment group from performing such a hierarchical comparison.
Time Frame: Up to 84 weeks
Population: Full analysis set: All patients included in the double-blind phase to whom study treatment was assigned by randomization and at least 1 dose of study treatment was received.
Measure: Number; unit: Pairwise comparisons
Units Other Than Participants: Pairwise comparison
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Open-label Phase Sacubitril+ Valsartan
Number analyzed (Participants) | 233 | 233 | 0
Number analyzed (Pairwise comparison) | 54289 | 54289 | 0
Pairwise comparisons
  Time to CV death wins | 2170 | 1536 |
  Time to CV death ties | 50583 | 50583 |
  Number and times of HF hospitalizations during follow-up wins: number analyzed (Pairwise comparison) | 50583 | 50583 | 0
  Number and times of HF hospitalizations during follow-up wins | 6963 | 6357 |
  Number and times of HF hospitalizations during follow-up ties: number analyzed (Pairwise comparison) | 50583 | 50583 | 0
  Number and times of HF hospitalizations during follow-up ties | 37263 | 37263 |
  Number and times of urgent HF visits during follow-up wins: number analyzed (Pairwise comparison) | 37263 | 37263 | 0
  Number and times of urgent HF visits during follow-up wins | 930 | 572 |
  Number and times of urgent HF visits during follow-up ties: number analyzed (Pairwise comparison) | 37263 | 37263 | 0
  Number and times of urgent HF visits during follow-up ties | 35761 | 35761 |
  Time-averaged proportional change in NT-proBNP wins: number analyzed (Pairwise comparison) | 35761 | 35761 | 0
  Time-averaged proportional change in NT-proBNP wins | 9987 | 8343 |
  Time-averaged proportional change in NT-proBNP ties: number analyzed (Pairwise comparison) | 35761 | 35761 | 0
  Time-averaged proportional change in NT-proBNP ties | 17431 | 17431 |
  Overall wins | 20050 | 16808 |
  Overall ties | 17431 | 17431 |
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Test type: Superiority; p = 0.1578, unmatched pairwise win-ratio; Win Ratio = 1.193, 95% CI 2-sided [0.934 to 1.524] — A win ratio greater than 1 was in favor of sacubitril/valsartan arm

3. Secondary Outcome: EAC Adjudicated Recurrent Composite Events
Description: This endpoint calculated the cumulative number of the following composite events over time:
  * CV death
  * recurrent HF hospitalizations
  * recurrent urgent HF visits The time to these recurrent events was analyzed using the semi-parametric proportional rates model (abbreviated as LWYY model).
  The exposure-adjusted rate per 100 subject years (EAR) was calculated diving the total number of events by 100 subject years (total exposure up to event/censoring).
  The role of the Endpoint Adjudication Committee (EAC) was to ensure that all treatment outcomes were judged uniformly, using standard criteria and processes.
  Events that occurred in the double-blind treatment phase are included in the analysis.
Time Frame: Up to Week 84
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: events per 100 subject years
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Open-label Phase Sacubitril+ Valsartan
Number analyzed (Participants) | 233 | 233 | 0
events per 100 subject years | 63.519 [51.330 to 77.732] | 76.189 [63.010 to 91.310] |
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Test type: Superiority; p = 0.3563, LWYY model; rate ratio = 0.8346, 95% CI 2-sided [0.5684 to 1.2255] — A rate ratio < 1 indicates an effect in favor of LCZ696

4. Secondary Outcome: Total Number of Confirmed Incidences of a Composite Endpoint of Worsening Renal Function
Description: This endpoint calculated the incidences of a composite endpoint of worsening renal function defined as:
  * renal death (from adverse events data)
  * reaching end-stage renal disease (ESRD) (Sustained eGFR <15mL/min/m2, chronic dialysis, or renal transplant)
  * ≥ 50% decline in estimated glomerular filtration rate (eGFR) relative to baseline [using central laboratory measurements (scheduled or unscheduled visits)]
  The Investigator-reported AE and central laboratory data was used to identified event of interest in this secondary endpoint.
  Events that occurred in the randomized double-blind treatment phase were included in the analysis.
Time Frame: Up to Week 84
Population: as for outcome 2
Measure: Number; unit: events of worsening renal function
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Open-label Phase Sacubitril+ Valsartan
Number analyzed (Participants) | 233 | 233 | 0
events of worsening renal function | 34 | 46 |
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Test type: Superiority; p = 0.3155, negative binomial regression model; Rate ratio = 0.6249, 95% CI 2-sided [0.2496 to 1.5649]

5. Secondary Outcome: Proportional Change in NT-proBNP From Baseline to Week 8
Description: This endpoint intended to assess the effect of sacubitril/valsartan vs. valsartan on change in N-terminal pro-brain natriuretic peptide (NT-proBNP) from baseline to Week 8.
  NT-proBNP is a protein produced in large amounts by the heart when it is not working properly, as in heart failure.
  The change from baseline to Week 8 was expressed as the geometric mean of the ratio: Week 8/Baseline.
Time Frame: Baseline and Week 8
Population: Full analysis set: All patients to whom study treatment was assigned by randomization and at least 1 dose of study treatment was received. Patients with missing baseline NT-proBNP and/or missing data from Week 8 were not included in the this analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan
Number analyzed (Participants) | 155 | 172
Geometric mean ratio | 0.6778 [0.5882 to 0.7810] | 0.7275 [0.6359 to 0.8323]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Test type: Superiority; p = 0.4766, ANCOVA; ratio of the change = 0.9316, 95% CI 2-sided [0.7661 to 1.1329]

6. Secondary Outcome: Proportional Change From Baseline in Hs-Troponin at Weeks 4 and 8
Description: This endpoint intended to assess the effect of sacubitril/valsartan vs. valsartan on change from baseline in high sensitivity (hs)-Troponin at Weeks 4 and 8. Analysis was repeated for both the visits, Week 4 and Week 8 separately.
  Hs-Troponin-T is a biomarker that is released from the heart under stress or injury conditions.
  The change from baseline to Week 4 and Week 8 was expressed as the geometric mean of the ratio: Week 4 or Week 8/Baseline.
Time Frame: Baseline, Week 4 and Week 8
Population: Full analysis set: All patients to whom study treatment was assigned by randomization and at least 1 dose of study treatment was received. Patients with missing baseline hs-Troponin and/or missing data from both Weeks 4 and 8 were not included in the this analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan
Number analyzed (Participants) | 171 | 187
Geometric mean ratio
  Week 4 | 0.8124 [0.76 to 0.87] | 0.9826 [0.92 to 1.05]
  Week 8: number analyzed (Participants) | 154 | 187
  Week 8 | 0.7545 [0.70 to 0.81] | 0.9310 [0.87 to 1.00]
Statistical Analysis 1: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Week 4; Test type: Superiority; p < .0001, ANCOVA; ratio of the change = 0.8268, 95% CI 2-sided [0.76 to 0.91]
Statistical Analysis 2: Comparison: Sacubitril/Valsartan (LCZ696) vs Valsartan; Week 8; Test type: Superiority; p < .0001, ANCOVA; ratio of the change = 0.8103, 95% CI 2-sided [0.74 to 0.89]

7. Secondary Outcome: Dosing Levels and Discontinuations
Description: The dosing level has been summarized by treatment group and in-/out-of-hospital randomization status. The dose levels used were:
  Dose Level 1: 40 mg valsartan or 24/26 mg [50 mg] LCZ696, BID; Dose Level 2: 80 mg valsartan or 49/51 mg [100 mg] LCZ696, BID; Dose Level 3: 160 mg valsartan or 97/103 mg [200 mg] LCZ696, BID
  Patients counted as "Off Treatment" are those who prematurely permanently discontinued study treatment but continued with visits.
  Patients counted as "No Treatment" are those who permanently discontinued with both study treatment and study visits
Time Frame: Randomization, Week 8, Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Open-label Phase Sacubitril+ Valsartan
Number analyzed (Participants) | 233 | 233 | 0
Participants
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): number analyzed (Participants) | 162 | 162 | 0
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): Dose Level 1 | 133 | 130 |
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): Dose Level 2 | 29 | 32 |
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): Dose Level 3 | 0 | 0 |
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): No Treatment | 0 | 0 |
  Participants Randomized In-Hospital ; Timepoint: Randomization (initial dose): Off Treatment | 0 | 0 |
  Participants Randomized In-Hospital ; Timepoint: Week 8: number analyzed (Participants) | 136 | 134 | 0
  Participants Randomized In-Hospital ; Timepoint: Week 8: Dose Level 1 | 29 | 40 |
  Participants Randomized In-Hospital ; Timepoint: Week 8: Dose Level 2 | 22 | 23 |
  Participants Randomized In-Hospital ; Timepoint: Week 8: Dose Level 3 | 48 | 48 |
  Participants Randomized In-Hospital ; Timepoint: Week 8: No Treatment | 27 | 18 |
  Participants Randomized In-Hospital ; Timepoint: Week 8: Off Treatment | 10 | 5 |
  Participants Randomized In-Hospital ; Timepoint: Week 24: number analyzed (Participants) | 71 | 78 | 0
  Participants Randomized In-Hospital ; Timepoint: Week 24: Dose Level 1 | 12 | 18 |
  Participants Randomized In-Hospital ; Timepoint: Week 24: Dose Level 2 | 5 | 16 |
  Participants Randomized In-Hospital ; Timepoint: Week 24: Dose Level 3 | 32 | 32 |
  Participants Randomized In-Hospital ; Timepoint: Week 24: No Treatment | 19 | 11 |
  Participants Randomized In-Hospital ; Timepoint: Week 24: Off Treatment | 3 | 1 |
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): number analyzed (Participants) | 71 | 71 | 0
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): Dose Level 1 | 62 | 60 |
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): Dose Level 2 | 9 | 11 |
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): Dose Level 3 | 0 | 0 |
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): No Treatment | 0 | 0 |
  Participants Randomized Out-of-hospital; Timepoint: Randomization (Initial Dose): Off Treatment | 0 | 0 |
  Participants Randomized Out-of-hospital; Timepoint: Week 8: number analyzed (Participants) | 60 | 59 | 0
  Participants Randomized Out-of-hospital; Timepoint: Week 8: Dose Level 1 | 18 | 21 |
  Participants Randomized Out-of-hospital; Timepoint: Week 8: Dose Level 2 | 15 | 12 |
  Participants Randomized Out-of-hospital; Timepoint: Week 8: Dose Level 3 | 22 | 20 |
  Participants Randomized Out-of-hospital; Timepoint: Week 8: No Treatment | 3 | 5 |
  Participants Randomized Out-of-hospital; Timepoint: Week 8: Off Treatment | 2 | 1 |
  Participants Randomized Out-of-hospital; Timepoint: Week 24: number analyzed (Participants) | 38 | 49 | 0
  Participants Randomized Out-of-hospital; Timepoint: Week 24: Dose Level 1 | 10 | 11 |
  Participants Randomized Out-of-hospital; Timepoint: Week 24: Dose Level 2 | 8 | 10 |
  Participants Randomized Out-of-hospital; Timepoint: Week 24: Dose Level 3 | 16 | 15 |
  Participants Randomized Out-of-hospital; Timepoint: Week 24: No Treatment | 3 | 9 |
  Participants Randomized Out-of-hospital; Timepoint: Week 24: Off Treatment | 1 | 4 |

8. Secondary Outcome: Incidence of Adverse Events of Special Interest (AESI) During Treatment
Description: This endpoint intended to calculate the incidence of the following adverse events of special interest (AESI) during treatment:
  Symptomatic hypotension, Hyperkalemia (potassium > 5.5 mEq/L), Angioedema and worsening renal function (defined as an increase in serum creatinine of ≥ 0.5 mg/dL and worsening of the eGFR by at least 25%)
Time Frame: Up to week 84
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sacubitril/Valsartan (LCZ696) | Valsartan | Open-label Phase Sacubitril+ Valsartan
Number analyzed (Participants) | 233 | 233 | 0
Participants
  Symptomatic hypotension | 56 | 36 |
  Hyperkalemia | 45 | 43 |
  Angioedema | 0 | 1 |
  Worsening renal function | 50 | 72 |

ADVERSE EVENTS:
Time Frame: Adverse events of the double-blind phase were reported from first dose of study treatment until end of study treatment plus 1 month post treatment, up to a maximum duration of 21 months. For those patients enrolled during the original version (00) of the protocol, where the open-label phase existed, adverse events were reported during the 4 week Open-Label period, and 1 month post treatment, for a maximum of 2 months.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Adverse events are provided by arm and not by dose as it was not planned in the analysis to provide AEs by dose.
Arm/Group | Double-blind Phase Sacubitril+ Valsartan (LCZ696) | Double-blind Phase Valsartan | Open-label Phase Sacubitril+ Valsartan
All-Cause Mortality (participants affected / at risk) | 18/233 | 26/233 | 0/50
Serious Adverse Events (participants affected / at risk) | 119/233 | 117/233 | 3/50
Other Adverse Events (participants affected / at risk) | 161/233 | 165/233 | 14/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase Sacubitril+ Valsartan (LCZ696) (N=233) | Double-blind Phase Valsartan (N=233) | Open-label Phase Sacubitril+ Valsartan (N=50)
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 5 | 4 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 8 | 0
Angina unstable (Cardiac disorders) | 0 | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 13 | 0
Atrial flutter (Cardiac disorders) | 1 | 2 | 0
Atrial tachycardia (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
BRASH syndrome (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac amyloidosis (Cardiac disorders) | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 4 | 3 | 0
Cardiac failure (Cardiac disorders) | 22 | 20 | 0
Cardiac failure acute (Cardiac disorders) | 11 | 14 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 14 | 19 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 2 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 4 | 1
Coronary artery disease (Cardiac disorders) | 3 | 4 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 2 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 1 | 5 | 0
Death (General disorders) | 6 | 7 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cyst ruptured (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Primary amyloidosis (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
COVID-19 (Infections and infestations) | 6 | 5 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 4 | 0
Cellulitis (Infections and infestations) | 1 | 6 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Histoplasmosis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 14 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 5 | 5 | 0
Septic shock (Infections and infestations) | 1 | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Wound infection bacterial (Infections and infestations) | 0 | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 4 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 2 | 0
Troponin increased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 4 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 2 | 0
Presyncope (Nervous system disorders) | 2 | 2 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 10 | 9 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 2 | 0
Device malfunction (Product Issues) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 21 | 15 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 4 | 3 | 0
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Dialysis hypotension (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Hypertensive emergency (Vascular disorders) | 0 | 4 | 0
Hypertensive urgency (Vascular disorders) | 1 | 3 | 0
Hypotension (Vascular disorders) | 15 | 13 | 0
Hypovolaemic shock (Vascular disorders) | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase Sacubitril+ Valsartan (LCZ696) (N=233) | Double-blind Phase Valsartan (N=233) | Open-label Phase Sacubitril+ Valsartan (N=50)
Atrial fibrillation (Cardiac disorders) | 9 | 13 | 1
Cardiac failure (Cardiac disorders) | 16 | 16 | 2
Constipation (Gastrointestinal disorders) | 6 | 12 | 0
Fatigue (General disorders) | 4 | 12 | 0
COVID-19 (Infections and infestations) | 18 | 14 | 0
Urinary tract infection (Infections and infestations) | 19 | 21 | 2
Fall (Injury, poisoning and procedural complications) | 16 | 14 | 0
Blood creatinine increased (Investigations) | 23 | 27 | 3
Glomerular filtration rate decreased (Investigations) | 4 | 4 | 3
SARS-CoV-2 test negative (Investigations) | 58 | 73 | 0
SARS-CoV-2 test positive (Investigations) | 23 | 18 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 38 | 43 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 22 | 1
Dizziness (Nervous system disorders) | 21 | 18 | 1
Acute kidney injury (Renal and urinary disorders) | 35 | 47 | 0
Chronic kidney disease (Renal and urinary disorders) | 6 | 15 | 1
Renal impairment (Renal and urinary disorders) | 11 | 20 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 1
Hypertension (Vascular disorders) | 8 | 12 | 0
Hypotension (Vascular disorders) | 58 | 40 | 1

LIMITATIONS AND CAVEATS:
No efficacy analyses include "OPEN LABEL' data. After Protocol Amendment 01, the open-label option was removed from the study, only the 233 patients randomized in the Double-blind Phase Sacubitril+ Valsartan (LCZ696) and the 233 patients randomized in the Double-blind Phase Valsartan arms were included in the efficacy analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03988634/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03988634/SAP_001.pdf